CLINICAL TRIAL: NCT05143749
Title: The Effects of Video Use and Self-evaluation on Gynecological Surgery Education in the Light of Current Technological Developments in the Pandemic
Brief Title: Pandemic and Gynecological Surgery Education
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: technical support not available
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Rahime Bedir Fındık, Associate Professor Dr, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AnkaraCHBilkent-MH-RBF-03
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Self Confidence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 assistant doctors who received video training (Experimental): 10 assistant doctors who receive video training will be the intervention arm
  Interventions: Other: video tutorial
- 10 assistant doctors who did not receive video training (No Intervention): 10 assistant doctors who did not receive video training will be the control arm

INTERVENTIONS:
Other: video tutorial — get video tutorial
  Arms: 10 assistant doctors who received video training

SUMMARY:
SarsCov2/COVID19 virus emerged in Wuhan, China in December 2019, and cases were seen in our country about 3 months later, causing a worldwide pandemic. In this process, both the stress caused by the risk of contracting the disease and the social restrictions affected life deeply.

578 / 5000 Çeviri sonuçları This study will be beneficial for the assistant doctors in recognizing technical errors in gynecological operations, reducing the risks and improving the results.

Surgical operation trainings such as hysterectomy and oophorectomy fistula surgery can be given with laparotomy-guided simulators, which can offer interactive training for gynecological operations in adult female sizes and show high adaptability. However, it is not possible to train major vaginal surgical operations with this method today. At this point, video tutorials can be used. This study was planned with the aim of increasing the level of anxiety about the training of the residents during the pandemic period, with the aim of making positive changes in order to increase the assistant's own skills, realize his mistakes and reduce the level of anxiety with video training.

DETAILED DESCRIPTION:
Our study is a Prospective Cross-sectional Case Control study. Our study is a training study and our assistants included in the study will consist of two groups. Group 1: A total of 10 assistants who have just completed the gynecological surgery training, which is in the last 4 months of a total of 8 months of training during the pandemic process, and Group 2 is 4 . It will consist of 10 assistants who have just started their surgical training after the first month. The assistants in Group 2 will videotape their first, fifth, tenth, fifteenth and twentieth gynecological operations, then watch their own operations to test their skills. Written consent will be obtained from the patients for the video recording of the operations, stating that the operations will be used for educational purposes only before the operation.

Operations are planned as abdominal hysterectomy, vaginal hysterectomy and myomectomy, which are the most performed gynecological operations.

Video applied to the residents in Group 1, who completed their training in the last 4 months of the pandemic process, and to the residents in Group 2, who completed their training by watching the video footage of their own operations, by applying the Self-Confidence Scale, General Self-Efficacy Scale, State Anxiety Inventory (DCI) and Trait Anxiety Inventory (SCI) scales. The effect of education on residents' anxiety, competence and self-confidence will be investigated.

After the training, the operations performed by the residents will be analyzed and the average operation time, intraoperative and postoperative major and minor complication rates, bleeding amounts in the operations, preoperative and postoperative hemogram amounts, postoperative hospital stay of the patients, postoperative analgesia need parameters will be evaluated and a comparison will be made between the two groups. In this way, the effect of video training on the lurning curve will be investigated.

ELIGIBILITY:
Inclusion Criteria: training as a gynecological assistant -

Exclusion Criteria:not yet receive gynecological assistant training

-

Ages: 24 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
self confidence | minimum 3 months
  Self-confidence level will be tested in the group receiving video training.

CONTACTS AND LOCATIONS:
Overall Officials: Rahime Bedir Findik, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No